CLINICAL TRIAL: NCT00147888
Title: Physiological Changes in Nasal Patency in Response to Changes in Posture, Temperature, Humidity and Nasal Patency Measured by Acoustic Rhinometry
Brief Title: Changes in Nasal Patency With Changes in Posture, Temperature, Humidity and Nasal Patency Seen by Acoustic Rhinometry
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13028A
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Mucosal Congestion
Keywords: Mucosal congestion; Acoustic rhinometry; Physiology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Acoustic rhinometry (procedure) — Acoustic rhinometry is a procedure that uses sound waves to measure the cross-sectional area and volume of the nasal cavity.

SUMMARY:
To study nasal physiologic responses to changes in posture, temperatures, humidity and nasal patency with acoustic rhinometry.

DETAILED DESCRIPTION:
The purpose of this study was to utilize acoustic rhinometry to assess changes in nasal patency after alterations in posture, unilateral mechanical obstruction, temperature, and humidity.

Eight healthy adult volunteer subjects underwent acoustic rhinometry under the following conditions: 1) upright, sitting position (control), 2) supine position, 3) left lateral recumbent position, 4) one nostril mechanically blocked, 5) icepack on neck, 6) drinking cold water, 7) drinking hot water, 8) nasal nebulizer, 9)oxymetazoline decongestant.

Changes in nasal cavity volumes were detected by acoustic rhinometry after alterations in posture, unilateral mechanical obstruction, temperature, and humidity. Nebulizer treatment and hot water ingestion caused a significant decrease in nasal volume. The nose was able to adapt to environmental and physiological changes in order to maintain a consistent total nasal volume.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, 18-58 years old

Exclusion Criteria:

* Any nasal symptoms in the last 3 weeks
* Marked septal deviation/polyposis/infection
* Any history of allergy, asthma or immunodeficiency
* Any systemic condition or infection (e.g., hypertension/diabetes/heart, liver, thyroid or kidney disease
* Any spine or neck condition that would not allow normal postures
* Pregnancy

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2004-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Changes in nasal patency | 5-10 minutes

SECONDARY OUTCOMES:
Nasal volume | 5-10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jacquelynne P. Corey, M.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Lundqvist GR, Pedersen OF, Hilberg O, Nielsen B. Nasal reaction to changes in whole body temperature. Acta Otolaryngol. 1993 Nov;113(6):783-8. doi: 10.3109/00016489309135901. PMID 8291439
- [Background] Yamagiwa M, Hilberg O, Pedersen OF, Lundqvist GR. Evaluation of the effect of localized skin cooling on nasal airway volume by acoustic rhinometry. Am Rev Respir Dis. 1990 Apr;141(4 Pt 1):1050-4. doi: 10.1164/ajrccm/141.4_Pt_1.1050. PMID 2327639
- [Background] DRETTNER B. VASCULAR REACTIONS ON THE INTAKE OF FOOD AND DRINK OF VARIOUS TEMPERATURES. Acta Otolaryngol Suppl. 1964;188:SUPPL 188:249+. doi: 10.3109/00016486409134570. No abstract available. PMID 14147452
- [Background] Kase Y, Hilberg O, Pedersen OF. Posture and nasal patency: evaluation by acoustic rhinometry. Acta Otolaryngol. 1994 Jan;114(1):70-4. doi: 10.3109/00016489409126019. PMID 8128857
- [Background] Fouke JM, Jackson AC. Acoustic rhinometry: effects of decongestants and posture on nasal patency. J Lab Clin Med. 1992 Apr;119(4):371-6. PMID 1583387
- [Background] Moinuddin R, Mamikoglu B, Barkatullah S, Corey JP. Detection of the nasal cycle. Am J Rhinol. 2001 Jan-Feb;15(1):35-9. doi: 10.2500/105065801781329473. PMID 11258653
- [Background] Haight JJ, Cole P. Reciprocating nasal airflow resistances. Acta Otolaryngol. 1984 Jan-Feb;97(1-2):93-8. doi: 10.3109/00016488409130968. PMID 6689832
- [Background] Hasegawa M. Nasal cycle and postural variations in nasal resistance. Ann Otol Rhinol Laryngol. 1982 Jan-Feb;91(1 Pt 1):112-4. doi: 10.1177/000348948209100125. No abstract available. PMID 7073167
- [Background] Rundcrantz H. Postural variations of nasal patency. Acta Otolaryngol. 1969 Nov;68(5):435-43. doi: 10.3109/00016486909121582. No abstract available. PMID 5378632
- [Background] Bickford L, Shakib S, Taverner D. The nasal airways response in normal subjects to oxymetazoline spray: randomized double-blind placebo-controlled trial. Br J Clin Pharmacol. 1999 Jul;48(1):53-6. doi: 10.1046/j.1365-2125.1999.00972.x. PMID 10383560
- [Background] Mamikoglu B, Houser S, Akbar I, Ng B, Corey JP. Acoustic rhinometry and computed tomography scans for the diagnosis of nasal septal deviation, with clinical correlation. Otolaryngol Head Neck Surg. 2000 Jul;123(1 Pt 1):61-8. doi: 10.1067/mhn.2000.105255. PMID 10889483
- [Background] Corey JP, Gungor A, Nelson R, Fredberg J, Lai V. A comparison of the nasal cross-sectional areas and volumes obtained with acoustic rhinometry and magnetic resonance imaging. Otolaryngol Head Neck Surg. 1997 Oct;117(4):349-54. doi: 10.1016/S0194-5998(97)70125-6. PMID 9339795
- [Background] Corey JP, Nalbone VP, Ng BA. Anatomic correlates of acoustic rhinometry as measured by rigid nasal endoscopy. Otolaryngol Head Neck Surg. 1999 Nov;121(5):572-6. doi: 10.1016/S0194-5998(99)70058-6. PMID 10547472
- [Background] Hendley JO, Abbott RD, Beasley PP, Gwaltney JM Jr. Effect of inhalation of hot humidified air on experimental rhinovirus infection. JAMA. 1994 Apr 13;271(14):1112-3. PMID 8151855
- [Background] Forstall GJ, Macknin ML, Yen-Lieberman BR, Medendrop SV. Effect of inhaling heated vapor on symptoms of the common cold. JAMA. 1994 Apr 13;271(14):1109-11. PMID 8151854
- [Background] Witek TJ Jr, Canestrari DA, Hernandez JR, Miller RD, Yang JY, Riker DK. Superficial nasal mucosal blood flow and nasal patency following topical oxymetazoline hydrochloride. Ann Allergy. 1992 Feb;68(2):165-8. PMID 1739191
- [Background] Corey JP, Kemker BJ, Nelson R, Gungor A. Evaluation of the nasal cavity by acoustic rhinometry in normal and allergic subjects. Otolaryngol Head Neck Surg. 1997 Jul;117(1):22-8. doi: 10.1016/S0194-59989770201-8. PMID 9230318
- [Background] Mamikoglu B, Houser SM, Corey JP. An interpretation method for objective assessment of nasal congestion with acoustic rhinometry. Laryngoscope. 2002 May;112(5):926-9. doi: 10.1097/00005537-200205000-00027. PMID 12150630
- [Background] Taverner D, Bickford L, Shakib S, Tonkin A. Evaluation of the dose-response relationship for intra-nasal oxymetazoline hydrochloride in normal adults. Eur J Clin Pharmacol. 1999 Sep;55(7):509-13. doi: 10.1007/s002280050665. PMID 10501820